CLINICAL TRIAL: NCT02136862
Title: A Natural History Study to Observe Disease Progression, Standard of Care and Investigate Biomarkers in Alport Syndrome Patients
Brief Title: ATHENA: Natural History of Disease Study in Alport Syndrome Patients
Acronym: RG012-01
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: RG012-01
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Alport Syndrome Patients With eGFR Between 45-90 ml/Min/1.73 m2
Keywords: Alport syndrome; kidney disease
MeSH Terms: conditions — Nephritis, Hereditary; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is limited published clinical data about the natural history of renal disease in Alport syndrome. The RG012-01 study will collect data to characterize the progression of renal dysfunction in Alport syndrome patients.

Patients with a confirmed diagnosis of Alport syndrome who have qualifying GFR will be considered for enrollment. The sequential sampling of subjects' urine and/or blood will allow an assessment of the rate of change of established clinical endpoints, such as GFR and/or the rate of change of other renal biomarkers (proteinuria and β-2 microglobulin) in subjects whose renal function is steadily declining. The identification of surrogate markers that track the decline of renal function and could correlate with time to end-stage renal disease (ESRD) is a key goal of the natural history study.

DETAILED DESCRIPTION:
This is a natural history study, designed to collect data from patients with Alport syndrome with qualifying GFR. Assessments and blood and urine sample collection will be performed at Baseline and every 12 weeks thereafter, for up to 120 weeks. Scheduling of clinic visits will take in to consideration the timing of Standard of Care (SOC) visits. Alternative arrangements may be made to enable subjects to schedule a home nurse visit for study procedures instead of certain clinic visits. Remaining blood and urine aliquots will be stored and may be used in the future for the discovery, analysis, verification and/or validation of other biomarkers or test for renal disease. The samples will be kept for up to five years. Each sample will be identified only by it's barcode number and will not be individually identifiable.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with the requirements of the study and willing and able to provide written informed consent; pediatric subjects must be able to provide assent;
* Age 12-65 years of age;
* Confirmed diagnosis of Alport syndrome (clinical, histopathologic and/or genetic diagnosis of Alport syndrome);
* eGFR 45-90 ml/min/1.73 m2, within 30 days of enrollment.

Exclusion Criteria:

* Use of investigational drugs at the time of enrollment, or within 30 days, or 5 half-lives of enrollment, whichever is longer;
* Ongoing chronic hemodialysis therapy and/or renal transplant recipient.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alport syndrome patients with eGFR between 45-90 ml/min/1.73 m2
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
To characterize the natural decline of renal function markers (Glomerular Filtration Rate [GFR] and creatinine) in patients with Alport syndrome over the course of up to 120 weeks | Up to 120 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director
Locations (15):
- United States (8):
  - San Diego, California
  - Chicago, Illinois
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Cleveland, Ohio
  - Plano, Texas
  - Salt Lake City, Utah
- Australia (2):
  - New Lambton, New South Wales
  - Parkville, Victoria
- Canada (2):
  - Vancouver, British Columbia
  - Toronto, Ontario
- Paris, France
- Göttingen, Germany
- London, United Kingdom